CLINICAL TRIAL: NCT06199791
Title: Single-Dose, Randomized, Two-Way Crossover, Bioequivalence of Lamotrigine 100 mg Tablet (Desitin Arzneimittel GmbH, Germany) and Lamictal 100 mg Tablet (GlaxoSmithKline GmbH & Co. KG, Germany) in Healthy, Male Volunteers, Fasting
Brief Title: Single-dose, Two-way Crossover Bioequivalence of Lamotrigine in Healthy Male Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Desitin Arzneimittel GmbH (Industry)
Collaborators: BioPharma Services Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LTG-008/K
Record Dates: First submitted 2023-12-12; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lamotrigine 100 mg oral tablet (Experimental): Test
  Interventions: Drug: Lamotrigine 100 MG
- Lamictal 100 mg oral tablet (Active Comparator): Reference
  Interventions: Drug: Lamotrigine 100 MG

INTERVENTIONS:
Drug: Lamotrigine 100 MG — tablets
  Other Names: Lamotrigin Desitin 100 mg

SUMMARY:
To assess the bioequivalence of lamotrigine from Lamotrigin Desitin 100 mg tablets and Lamictal 100 mg Tablet.

DETAILED DESCRIPTION:
In the pivotal study bioequivalence of Lamotrigin Desitin 100 mg tablets and Lamictal 100 mg tablet in healthy, male volunteers should be proven.

The drug products were studied using a crossover design with 24 healthy, non-smoking, male volunteers being administered an oral dose of 1 × 100 mg tablet under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking (for at least 6 months prior to first drug administration), male volunteers 18 to 65 years of age inclusive.
2. BMI that was within 18.5-30.0 kg/m², inclusive.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
4. QTcB interval < 440 milliseconds for males, unless deemed otherwise by the PI/Sub- Investigator.
5. Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
6. Clinical laboratory values within BPSI's most recent acceptable laboratory test range, and/or values were deemed by the PI/Sub-Investigator as "Not Clinically Significant".
7. Ability to comprehend and be informed of the nature of the study, as assessed by BPSI staff. Capable of giving written informed consent prior to any study-related procedure.

   Must have been able to communicate effectively with clinic staff.
8. Ability to fast for at least 14 hours and consume standard meals.
9. Availability to volunteer for the entire study duration and was willing to adhere to all protocol requirements.
10. Agreed not to have a tattoo or body piercing until the end of the study.
11. Agreed not to receive the COVID-19 vaccination from 7 days prior to the first study drug dose until 7 days after the last study drug administration in the study.
12. Agreed to limit exposure to sunlight and UV light by wearing protective clothing and using a sunscreen with a high protection factor during the study.
13. Agreed not to drive or operate heavy machinery if feeling dizzy or drowsy following study drug administration until full mental alertness was regained.
14. Males who were able to father children agreed to use medically acceptable methods of contraception during the study and for 30 days after the last study drug administration.

Medically acceptable methods of contraception included using a condom with a female partner of child-bearing potential who was using oral contraceptives, hormonal patch, implant or injection, intrauterine device, or diaphragm with spermicide. Abstinence as a method of contraception was acceptable if it was in line with the preferred and usual lifestyle of the study participant. If a subject's partner became pregnant during his participation in the study and for 30 days after he had completed his last study drug administration, he must have informed BPSI staff immediately.

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.
3. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
4. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
5. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol breath test and cotinine.
6. Known history or presence of:

   * Alcohol abuse or dependence within one year prior to first study drug administration.
   * Drug abuse or dependence within the last 2 years.
   * Prior history or family history of hypersensitivity or idiosyncratic reaction to any drug including but not limited to Lamotrigine, its excipients, and/or related substances;
   * Suicidal ideation or suicidal behavior, as assessed by the Columbia Suicide Severity Rating Scale (baseline version) - Appendix B (Refer to Appendix 16.1.1)
   * Prior history or family history of allergic drug rash to any drug including but not limited to lamotrigine, its inactive ingredients and/or any other related marketed drugs, including Lamictal XR and Lamictal.
   * Prior history or family history of Stevens-Johnson Syndrome (SJS);
   * Lactose intolerance;
   * Food allergies;
   * Presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant".
   * Severe allergic reactions (e.g., anaphylactic reactions, angioedema).
7. Intolerance to and/or difficulty with blood sampling through venipuncture.
8. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets etc.
9. Individuals who had donated, in the days prior to first study drug administration:

   * 50-499 mL of blood in the previous 30 days;
   * 500 mL or more in the previous 56 days.
10. Donated plasma by plasmapheresis within 7 days prior to first study drug administration.
11. Individuals who had participated in another clinical trial or who received an investigational drug within 30 days prior to first study drug administration.
12. Use of any enzyme-modifying drugs and/or other products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort, and rifampicin) in the previous 30 days before first study drug administration.
13. Used any prescription medication within 14 days prior to first study drug administration (except for spermicidal/barrier contraceptive products).
14. Used of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 14 days prior to first study drug administration (except for spermicidal/barrier contraceptive products).
15. Used Acetaminophen (Paracetamol) during the study.
16. Consumed food or beverages containing grapefruit and/or pomelo within 10 days prior to first study drug administration.
17. Consumed food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing in each study period.
18. Individuals who had undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.
19. Difficulty with swallowing whole tablet.
20. Unable or unwilling to provide informed consent.
21. Had a tattoo or body piercing within 30 days prior to first study drug administration.
22. Recent history (within 8 weeks prior to screening) of travel to or emigration from any country with high incidence for tuberculosis.
23. History or presence of tuberculosis or a positive QUANTIFERON blood test/Tuberculin Skin Test result.
24. A subject who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | blood sampling: pre-dose (0) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose
  To establish bioequivalence, the calculated 90% CI for the ratio of geometric means for AUC72 and Cmax for lamotrigine should fall within 80.00%-125.00%.
Maximal plasma concentration (Cmax) | blood sampling: pre-dose (0) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose
  To establish bioequivalence, the calculated 90% CI for the ratio of geometric means for AUC72 and Cmax for lamotrigine should fall within 80.00%-125.00%.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Faulknor, MD, Principal Investigator — BioPharma Services Inc.
Locations (1):
- Biopharma Services INC, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No